CLINICAL TRIAL: NCT03081468
Title: A Prospective Single-Site Non-Interventional Study to Evaluate the Diagnostic Accuracy and Repeatability of Pupil Measurements Using a Prototype Binocular Optical Coherence Tomography System.
Brief Title: The PUPIL Study - Automated, Quantitative Pupil Assessment Using Binocular OCT
Status: Completed | Type: Observational
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 16/0578
Record Dates: First submitted 2017-03-10; First posted 2017-03-16 (Actual); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Healthy Volunteers; Relative Afferent Pupil Defect; Pupil Anomaly
Keywords: Optical coherence tomography; Pupillometry; Automated; Binocular
MeSH Terms: conditions — Pupil Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy volunteers: Fifty healthy volunteers. Each participant will attend for a single study visit, lasting approximately 1 hour in duration. Participants will undergo pupillometry examination using the binocular OCT prototype and Konan RAPDx.
  Interventions: Device: Binocular OCT prototype; Device: Konan RAPDx
- Participants with confirmed relative afferent pupillary defect: Fifty participants with with eye disease (retinal disease, glaucoma, and neuro-ophthalmic conditions) and confirmed relative afferent pupillary defect. Each participant will attend for a single study visit, lasting approximately 1 hour in duration. Participants will undergo pupillometry examination using the binocular OCT prototype and Konan RAPDx.
  Interventions: Device: Binocular OCT prototype; Device: Konan RAPDx

INTERVENTIONS:
Device: Binocular OCT prototype — Participants in the study will undergo pupil measurement using a prototype binocular OCT imaging system (Envision Diagnostics, Inc., CA). For the binocular OCT imaging system, testing will be performed twice in the same session, by the same examiner, to allow assessment of repeatability (test-retest variability).
Device: Konan RAPDx — Participants in the study will undergo pupil measurement using a validated, commercially available pupilometer (RAPDx; Konan Medical USA, Inc., Irvine, CA).

SUMMARY:
In current, clinical ophthalmology, a range of specialised testing allows comprehensive evaluation of ocular health. These tests have typically evolved over many years to ensure their clinical validity. For example, the assessment of visual acuity has traditionally been measured with Snellen letter charts from a distance of six metres (20 feet), leading to the phrase "20/20 vision". Despite this, the limitations of Snellen testing are well established and more sophisticated testing is now available (e.g., logMAR testing using ETDRS (Early Treatment Diabetic Retinopathy Study) charts). Many other diagnostic tests have undergone similar cycles of refinement, often over extended time periods. Therefore, it should be incumbent on any new device to undergo detailed evaluation of its validity (how its measurements agree with other testing) and its repeatability (the variability when a further measurement is obtained in short time period, by the same operator and under the same conditions).

Binocular OCT extends the application of OCT devices beyond that of simple, cross- sectional imaging to a diverse array of diagnostic tests. The binocular design also removes the need for additional personnel to perform testing (i.e., the device can be self-operated in an automated manner), and allows for novel testing to be performed that is not possible with monocular imaging. In particular, binocular OCT devices have the potential to perform automated, quantitative pupillary measurements - an entirely novel application for this imaging modality.

This study will assess the validity and repeatability of pupil measurements using binocular OCT.

DETAILED DESCRIPTION:
Binocular OCT has the potential to allow for objective, quantitative measurement of pupillary reflexes, that can be performed in a fast, safe, and automated manner. Importantly, binocular OCT pupillometry can be performed alongside binocular retinal OCT imaging in a single testing session, in an automated manner (imaging of the retina using OCT is the commonest ophthalmic imaging procedure worldwide - in 2011, it is estimated that more than 20 million retinal OCT images were obtained, more than the sum of all other ophthalmic imaging procedures combined).

Assessment of pupillary reflexes is an essential component of a comprehensive ocular examination. In patients with visual loss, for example, detection of an RAPD often indicates the presence of serious ophthalmic diseases, such as optic neuropathies or severe retinal disease. As such, RAPD testing is essential as a screening test in the assessment of patients with less serious conditions such as cataract.

RAPD testing is commonly performed using the swinging flashlight method (SFM). A positive SFM test suggests the presence of asymmetric damage involving the afferent limb of the pupillary light reflex pathway. The SFM is a qualitative test, and relies upon visualising no pupillary constriction or immediate or delayed pupillary dilation; if either of these responses is observed, an RAPD is believed to be present. The SFM requires a trained examiner and many potential sources of error may confound the results, including anisocoria, off-axis pupil illumination, and unequal retinal bleaching. Pupil abnormalities may be subtle and easily missed using the SFM.

Automated pupilometers allow examiners to precisely and objectively quantify the pupillary response to light by measuring parameters such as minimum and maximum pupil diameter, the amplitude of constriction, latency of constriction, velocity of constriction, and duration of maximum constriction. Dedicated pupillometry devices are commercially available and have been shown to be highly sensitive and specific for RAPD detection e.g. RAPDx; Konan Medical USA, Inc., Irvine, CA. These devices are also capable of detecting the presence of more subtle RAPD, typically not found using the SFM, in diseases such as glaucoma.

Unfortunately, automated pupilometers such as the Konan RAPDx system are not widely used in clinical practice. This is largely because they are expensive devices, limited to a single purpose. A binocular OCT system that could perform both automated pupillometry and retinal OCT imaging would thus have great clinical utility.

ELIGIBILITY:
Inclusion criteria for participants with eye disease will include:

* Presence of RAPD as measured with RAPDx
* Presence of retinal disease, glaucoma or neuro-ophthalmic conditions that affect the optic nerve
* Male or female, aged 18 years or older
* Ability to understand nature/purpose of the study and to provide informed consent
* Ability to undergo binocular OCT imaging
* Ability to follow instructions and complete the study
* Ability to speak English

Exclusion criteria for participants with eye disease will include:

* Optical media opacity sufficient to preclude adequate ocular imaging with OCT
* Ptosis (drooping of the upper eyelid) sufficient to preclude visualization of the pupils using OCT
* Significant pupil irregularity that precludes reliable measurement of RAPD
* Any condition that is likely to interfere with pupillary constriction (e.g., iris pathology)
* Hearing impairment sufficient to interfere with hearing instructions
* Any condition which, in the investigator's opinion, would conflict or otherwise prevent the subject from complying with the required procedures, schedule, or other study conduct.

Inclusion criteria for healthy subjects will include:

* No self-reported ocular history (although wearing corrective prescription glasses is permitted)
* Male or female, aged 18 years or older
* Ability to understand nature/purpose of the study and to provide informed consent
* Ability to undergo binocular OCT imaging
* Ability to follow instructions and complete the study
* Ability to speak English

Exclusion criteria for healthy subjects will include:

* Presence of ocular pathology, including ptosis or pupil irregularities
* Hearing impairment sufficient to interfere with hearing instructions
* Any condition which, in the investigator's opinion, would conflict or otherwise prevent the subject from complying with the required procedures, schedule, or other study conduct.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with eye disease (retinal disease, glaucoma, and neuro-ophthalmic conditions), and confirmed relative afferent pupillary defect as measured with RAPDx, and participants with no ocular abnormality ("healthy volunteers") will be recruited for the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-05-18 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of the binocular OCT | 6 months
  The primary objective will be to determine the diagnostic accuracy of a prototype binocular OCT system for the detection of relative afferent pupillary defect (RAPD).

SECONDARY OUTCOMES:
Test-retest variability of the binocular OCT pupillometry assessment | 6 months
  The secondary objective will be to assess the repeatability (test-retest variability) of pupillary assessment using this prototype binocular OCT system.

CONTACTS AND LOCATIONS:
Locations (1):
- Moorfields Eye Hospital NHS FT, London, United Kingdom